CLINICAL TRIAL: NCT00672646
Title: A Double-blind, Randomized, Placebo and Naproxen Controlled Study to Investigate the Analgesic Efficacy of a Single Dose of AZD1386, in Patients Undergoing Impacted Mandibular Third Molar Extraction
Brief Title: Study to Investigate the Analgesic Efficacy of a Single Dose of AZD1386
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D5090C00010
Record Dates: First submitted 2008-05-01; First posted 2008-05-06 (Estimated); Results first posted 2012-06-08 (Estimated); Last update posted 2012-06-08 (Estimated); Status verified 2012-05

CONDITIONS: Pain
Keywords: Analgesic effect
MeSH Terms: conditions — Pain | interventions — AZD1386; Naproxen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (3):
- AZD1386 (Experimental)
  Interventions: Drug: AZD1386
- Naproxen (Active Comparator)
  Interventions: Drug: Naproxen
- Placebo (Placebo Comparator): Placebo matching AZD1386
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD1386 — 95mg, oral solution, single dose
  Arms: AZD1386
Drug: Naproxen — 500mg, capsule, single dose
  Arms: Naproxen
Drug: Placebo — AZD1386 Placebo oral solution
  Arms: Placebo

SUMMARY:
The primary aim of this study is to investigate if AZD1386 can relieve the pain induced by the surgical removal of one lower wisdom-tooth. This will be done by comparing the effect of AZD1386 to placebo ("inactive substance") on pain. A number of patients will instead receive the common painkiller naproxen for comparison purposes. Rescue medication, acetaminophen, will be allowed if a need for additional painkillers would arise. A number of patients will receive naproxen as control.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for surgical removal of one partial or complete impacted mandibular third molar.
* Provision of signed informed consent.

Exclusion Criteria:

* History of somatic disease/condition, which may interfere with the objectives for the study, as judged by the investigator.
* Clinically significant illness or clinically relevant trauma within the 2 weeks prior to the administration of the investigational product, as judged by the investigator.
* A family history of short QT syndrome (SQTS) or sudden cardiac death (SCD) amongst first degree relatives
* Patients with a body temperature >37.5°C at Visit 2, before start of surgical procedures

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 103 (Actual)
Dates: Start 2008-04; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Webster, MD, Principal Investigator — Lifetree Clinical Research3838 South, 700 East, Suite 202Salt Lake City, Utah 84106, USA; Bror Jonzon, Study Chair — AstraZeneca R&D Södertälje, SE-151 85 Södertälje, Sweden
Locations (1):
- Research Site, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was performed at Lifetree Clinical Research, Salt Lake City, USA, during April-June 2008.
  135 participants enrolled in the study, 103 randomized and 99 patients completed the study.
Pre-assignment Details: Screening for eligibility prior to the residential day, and selecting the patients that request pain relief, due to pain from the dental surgical area, within 6 hours after the end of the administration of the local anaesthetic.
Groups:
- AZD1386: AZD1386 95 mg oral solution
- Naproxen: Naproxen 500 mg capsule
Period: Overall Study
Arm/Group | AZD1386 | Naproxen | Placebo
Started | 40 | 23 | 40
Completed | 40 | 22 | 37
Not Completed | 0 | 1 | 3
Not completed — Lost to Follow-up | 0 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD1386 | Naproxen | Placebo | Total
Number analyzed (Participants) | 40 | 23 | 40 | 103
Age Continuous [Mean (Standard Deviation); unit: year] | 21.5 (4.4) | 21 (4.8) | 21.9 (4.8) | 21.5 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 40 | 23 | 40 | 103

OUTCOME MEASURES:

1. Primary Outcome: Sum of Pain Intensity Difference in Percent (SPID%)
Description: Weighted sum of the pain intensity (PI) differences in percent for the given time frame. PI values are weighted according to the time since the previous PI assessment (or the time of administration of the investigational product for the first post-dose assessment). SPID% = elapsed since previous value, where is the PI difference in percent at assessment t. High values=good effect, low values=poor effect Pointwise assessments of pain are measured using a VAS scale (0-100 mm), as described in the secondary outcome measure (PI).
Time Frame: from the start of administration of the investigational product up to the time of first administration of rescue analgesic or up to a maximum of 8 hours
Measure: Median (Full Range); unit: percentage of pain intensity change * h
Arm/Group | AZD1386 | Naproxen | Placebo
Number analyzed (Participants) | 40 | 23 | 40
percentage of pain intensity change * h | 35.5 [-156.4 to 603.7] | 171.8 [-723.8 to 709.8] | -7.5 [-106.5 to 588.7]

2. Secondary Outcome: Pain Intensity (PI) by Using Visual Analogue Scale (VAS) (0-100 mm)
Description: 0 = 'No pain' 100 ='Worst pain imaginable' Up to 16 individual assessments were performed and contained in the derived primary outcome measure, thus not reported separately.
Time Frame: Immediately prior to administration of investigational product (IP). After intake of IP assessment will be made every 15 min for the first 2 h, at 2h and 30 min, 3 h and thereafter every hour up to 8 h after intake of IP.
Measure: Median (Full Range); unit: units on VAS scale
Arm/Group | AZD1386 | Naproxen | Placebo
Number analyzed (Participants) | 40 | 23 | 40
units on VAS scale
  Just before dosing | 50 [16 to 86] | 48 [13 to 90] | 46.5 [13 to 87]
  15 minutes | 33 [0 to 85] | 54 [9 to 89] | 45 [3 to 96]
  30 minutes | 30.5 [0 to 92] | 61 [17 to 90] | 47 [3 to 100]
  45 minutes | 28.5 [0 to 96] | 61 [12 to 89] | 51 [5 to 100]
  1 hour | 31.5 [1 to 84] | 52 [5 to 94] | 55 [7 to 100]
  1 hour 15 minutes | 35.5 [6 to 100] | 46 [3 to 86] | 53 [7 to 100]
  1 hour 30 minutes | 41 [8 to 100] | 38 [3 to 89] | 44 [4 to 100]
  1 hour 45 minutes | 50.5 [8 to 93] | 35 [1 to 70] | 50 [3 to 93]
  2 hours | 50.5 [9 to 91] | 28 [0 to 76] | 37 [1 to 79]
  2 hours 30 minutes | 30.5 [4 to 81] | 26 [0 to 79] | 23 [0 to 87]
  3 hours | 24.5 [0 to 71] | 21 [0 to 73] | 20 [0 to 92]
  4 hours | 14 [0 to 89] | 18 [0 to 70] | 14.5 [0 to 79]
  5 hours | 19 [0 to 83] | 10 [0 to 73] | 14 [0 to 51]
  6 hours | 14 [0 to 68] | 7 [0 to 68] | 13 [0 to 40]
  7 hours | 15 [0 to 55] | 6 [0 to 66] | 14 [0 to 44]
  8 hours | 14 [0 to 56] | 4 [0 to 73] | 11.5 [0 to 44]

3. Secondary Outcome: Time to First Perceptible Pain Relief
Description: First perceptible pain relief is the time at which the participant begins to feel any pain relief at all. The time to first perceptible pain relief was reported by the participant using a stopwatch. Each time the watch is stopped, the participants will rate their pain intensity. Note: Participants who do not report first perceptible pain relief, and participants who report first perceptible pain relief after rescue intake, have the corresponding time censored to 8 hours.
Time Frame: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: hour
Arm/Group | AZD1386 | Naproxen | Placebo
Number analyzed (Participants) | 40 | 23 | 40
hour | 0.3 [0.2 to 0.9] | 0.8 [0.4 to 4.2] | 1.3 [0.4 to 8]

4. Secondary Outcome: Time to First Meaningful Pain Relief
Description: First meaningful pain relief is the time when the participant's pain relief feels meaningful. The time to first meaningful pain relief will be reported by the participant using a stopwatch. Each time the watch is stopped, the participants will rate their pain intensity. Note: Participants who do not report first meaningful pain relief, and participants who report first meaningful pain relief after rescue intake, have the corresponding time censored to 8 hours.
Time Frame: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: hour
Arm/Group | AZD1386 | Naproxen | Placebo
Number analyzed (Participants) | 40 | 23 | 40
hour | 8.0 [0.9 to 8.0] | 4.2 [1.5 to 8.0] | 8.0 [6.5 to 8.0]

5. Secondary Outcome: VAS Pain Intensity at Rescue Intake
Description: 0 = 'No pain' 100 ='Worst pain imaginable'
Time Frame: at the time of first administration of rescue analgesic, up to the maximum time of 8 hours after intake of the investigational product
Population: Only participants that took rescue medication are included in this analysis.
Measure: Median (Full Range); unit: units on a VAS scale
Arm/Group | AZD1386 | Naproxen | Placebo
Number analyzed (Participants) | 32 | 11 | 32
units on a VAS scale | 61.0 [19.0 to 100.0] | 69.0 [26.0 to 93.0] | 70.5 [14.0 to 100.0]

6. Secondary Outcome: VAS Pain on Jaw Movement at Rescue Intake
Description: 0 = 'No pain' 100 ='Worst pain imaginable'
Time Frame: as for outcome 5
Population: Only participants that took rescue medication are included in this analysis.
Measure: Median (Full Range); unit: Units on a VAS scale
Arm/Group | AZD1386 | Naproxen | Placebo
Number analyzed (Participants) | 32 | 11 | 32
Units on a VAS scale | 65.0 [8.0 to 100.0] | 81.0 [16.0 to 96.0] | 73.5 [5.0 to 100.0]

ADVERSE EVENTS:
Arm/Group | AZD1386 | Naproxen | Placebo
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/23 | 0/40
Other Adverse Events (participants affected / at risk) | 4/40 | 0/23 | 6/40
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZD1386 (N=40) | Naproxen (N=23) | Placebo (N=40)
CHILLS (General disorders) | 2 | 0 | 0
DIZZINESS (Nervous system disorders) | 0 | 0 | 4
HEADACHE (Nervous system disorders) | 2 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AstraZeneca has the exclusive right to publish the results of the study.